CLINICAL TRIAL: NCT04219683
Title: Mandibular Vertical Height Augmentation in Segmental Defects Using Combined Vascularized and Non-Vascularized Fibula Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Magdy AbdelMoaz, Resident in Oral and Maxillofacial Surgery Department faculty of dentistry- Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-01-03
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Mandibular Reconstruction Using Free Fibula Flap
Keywords: free fibula flap - Mandibular reconstruction - Segmental Defects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with resected Mandible (Experimental): Patient with resected mandible who is candidate for free fibula flap
  Interventions: Procedure: Mandibular vertical height augmentation in segmental defects using combined vascularized and non-vascularized fibula flap

INTERVENTIONS:
Procedure: Mandibular vertical height augmentation in segmental defects using combined vascularized and non-vascularized fibula flap — Using Free Fibula Flap for reconstruction of mandibular segemental defect

SUMMARY:
Segmental mandibulectomy, often employed for resection of a tumour, and occasionally for trauma, osteoradionecrosis, or osteomyelitis, adversely affects patient's quality of life (QoL) to a varying degree. It inflicts a significant defect in the head and neck region, impacting on facial appearance, and the functions of speech, malocclusion, mastication, swallowing, and health-related QoL. Mandible resection thus creates a significant impact on a patient's life, both aesthetically as well as functionally.

Restoration of the defects following resection of any part of the mandible presents a challenging problem for reconstructive surgeons. Since the introduction of fibula free flap (FFF) by Taylor in 1975, it has become the most popular choice for mandible reconstruction. Hidalgo popularized the FFF, and reported on its versatility with satisfactory outcomes. The utility and techniques of free flap mandible reconstruction have advanced in the past 2 decades, with success rate up from 82.6% to 100%. As the longest bone segment available for reconstructive purpose, FFF is known for its wide variety of applications, following mandible resection, including angle-to-angle reconstruction.

The fibula-free flap is currently considered the most popular, 'the gold standard and the workhorse flap' for mandibular reconstruction.

However, because of the limited diameter of the fibula flap compared with the height of the mandible, vertical distance between the reconstructed segment and the occlusal plane can be substantial. This is a particular problem in the dentate mandible, especially when rehabilitation with dental implants or an implant-borne denture is contemplated. Insufficient bone height leads to overloading of osteointegrated implants and endangers the longevity of the prosthetic restoration. Insufficient bone height and poor soft tissue overlying the bone flap also create an unfavourable environment for the tissue-borne prosthesis.

Such issues are particularly acute in patients with intact alveolar bone and dentition at healthy sites. The double-barrel technique, distraction osteogenesis, non-vascularized bone grafts, and guided-bone regeneration have all been used to resolve this. The double-barrel technique is a good method, but drawbacks include excess height of the neomandible and the considerable time required to contour and adapt the upper barrel. Distraction osteogenesis is a valuable and predictable treatment option; however, its wide application is limited by complexity of the surgery and the need for additional secondary surgery.

To Overcome these challenges the investigators design a technique for mandibular reconstruction where free vascularized fibula flap is splitted and non-vascularized fibula graft is harvest from same leg and is placed between two splitted parts of free fibula flap to increase vertical height of fibula.

ELIGIBILITY:
Inclusion Criteria:

* Patient who require mandibular resection due to tumor, trauma, osteomyelitis or osteoradionecrosis.
* Patient with Mandibular defect >9 cm.

Exclusion Criteria:

* Patients with systemic condition counteracting with the surgical procedure.
* Patients with conditions contraindicating fibular flap.
* Patients with extensive defects of the mandible where the length of the harvested fibula flap would not allow for simultaneous ipsilateral harvesting of a non-vascularized segment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Height of mandible | one year
  Amount of vertical height gain (Mandibular augmentation) using Multi-slice CT Scan - Measured in millimeters

SECONDARY OUTCOMES:
Patient Satisfaction: Visual analogue Scale | One year
  Patient Satisfaction using Visual analogue Scale - Scale from 0-10